CLINICAL TRIAL: NCT04338295
Title: Follicular Revival in Treatment-resistant Alopecia Areata: Evaluating Use of Micro-needling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2000027352
Record Dates: First submitted 2020-04-03; First posted 2020-04-08 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Microneedling (Experimental): Participants with Alopecia Areata will receive microneedling with a tattoo machine.
  Interventions: Device: Tattoo machine (SOL Nova Device)

INTERVENTIONS:
Device: Tattoo machine (SOL Nova Device) — A SOL Nova Device (brand) tattoo machine will be used to stimulate hair regrowth.

SUMMARY:
The investigators propose to study the efficacy of micro-needling via the SOL Nova Device in generating hair growth in patients with Alopecia Areta (AA) who are either non-responsive or only partially responsive to combination oral JAK inhibitor plus oral minoxidil therapy.

DETAILED DESCRIPTION:
This will be a trial evaluating the efficacy of micro-needling via tattoo device in stimulating scalp hair growth in patients with AA refractory to combination JAK inhibitor and oral minoxidil treatment. Ten healthy subjects who are at least eighteen years of age who have experienced no or partial scalp hair regrowth after ≥three months of JAK inhibitor plus oral minoxidil treatment will be enrolled. Subjects will undergo a treatment session once every thirty days for a total of six sessions over six months and will complete a total of eight visits over eight months. Procedures and visits are not standard of care but conducted for research. Each visit will last about an hour. Approximately 30 minutes will be spent on consenting and time for patient to ask questions during the first visit. The remaining 30 minutes will be allotted for the investigator to determine if the patient meets criteria for trial enrollment. During the remaining visits, 20 minutes will be allotted for photography, 15-20 minutes for the procedure and 10-15 minutes for post-procedure patient assessment. Remaining 10 minutes on visits 2 and 8 will be used for biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AA
* SALT score ≥90%
* No or minimal scalp hair regrowth after ≥three months of oral JAK inhibitor plus oral minoxidil treatment

Exclusion Criteria:

* Known concomitant androgenetic or other form of alopecia (in addition to AA)
* Patients with the following who would make poor candidates for microneedling such as skin conditions, diabetes, or history of keloid formation
* Anything additional existing comorbidities that in the opinion of the investigator may cause unnecessary risk for the patient to participate

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-05-16 (Actual)

PRIMARY OUTCOMES:
Target area hair count (TAHC) | 6 months
  Total number of hairs in the area that undergoes microneedling

SECONDARY OUTCOMES:
Hair phase | 6 months
  Number of catagen, anagen hairs
Vellus hairs | 6 months
  Number of vellus hairs in an area of 1cm^2
Terminal hairs | 6 months
  Number of terminal hairs in an area of 1cm^2

CONTACTS AND LOCATIONS:
Overall Officials: Brett King, MD, PhD, Principal Investigator — Associate Professor of Dermatology, Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No